CLINICAL TRIAL: NCT06440291
Title: Effects of caRdioneurOablation on Exercise perforMance in Patients With Reflex Asystolic syNcope: The Roman 3 Study
Brief Title: Cardioneuroablation for Reflex Syncope and Exercise Capacity
Acronym: Roman3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, Professor, Centre of Postgraduate Medical Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 501-1-10-14-24
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Syncope, Vasovagal
Keywords: syncope
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cardioneuroablation (Experimental): Cardioneuroablation procedure as described in the Methods section of the study
  Interventions: Procedure: Cardioneuroablation

INTERVENTIONS:
Procedure: Cardioneuroablation — Cardioneuroablation procedure performed according to the protocol

SUMMARY:
Cardioneuroablation (CNA) is a new promising method to treat reflex syncope which is due to vagally-induced functional sinus arrest or atrio-ventricular block (AVB). Although the procedure is effective in > 80% of patients, there are potential adverse effects associated with the lack of vagal protection. One of them is increased sinus rate and possible worsening of exercise capacity. However, it is not known how often this happens. Moreover, the most accurate tool to asses exercise capacity - cardiopulmonary exercise testing (CPET), has not yet been used in this group of patients. Therefore, the aim of the study is to assess one-year effects of CNA-induced total vagal denervation on cardiorespiratory fitness in patients undergoing CNA due to reflex asystolic syncope.

The study group consists of patients undergoing CNA in our institution. All patients give informed written consent to undergo CNA and to participate in the study (Ethics Committee approval # 22/2024). CNA is performed according to standard protocol used in our institution. A symptom-limited cardiopulmonary exercise (CPET) is performed twice, at baseline (1-2 days before CNA) and after one year of follow-up. Standard CPET parameters are measured. Quality of life is measured using a dedicated questionnaire. Also, a control group of healthy volunteers will undergo CPET to answer the question whether subjects with reflex syncope differ in exercise capacity from healthy people.

DETAILED DESCRIPTION:
Introduction Cardioneuroablation (CNA) is a new promising method to treat reflex syncope which is due to vagally-induced functional sinus arrest or atrio-ventricular block (AVB). The goal of the procedure is to ablate post-ganglionic endings of the parasympathetic part of the autonomic nervous system (ANS), located in ganglionated plexi (GP) in the epicardial fat and in the myocardium. Although both sympathetic and parasympathetic nerves are localized in GPs, the latter ones only barely regenerate. Therefore, CNA-induced damage to the parasympathetic part of GP is greater and more durable than that of the sympathetic part of ANS. Because increased vagal activity is one of the main mechanisms leading to reflex sinus arrest or atrio-ventricular (AV) block, targeting this part of ANS by CNA may prevent recurrences of reflex syncope. Indeed, it has been shown that CNA may be effective in approximately 80-90% of very symptomatic subjects with reflex syncope.

Lack or diminished parasympathetic drive to the heart may be, however, associated with adverse effects. The main complication which is seen shortly and up to one year after CNA is heart rhythm acceleration which may be symptomatic in approximately one-third of patients. In the majority of patients sinus rate gradually slows down over a period of 3-12 months due to partial parasympathetic reinnervation, however, approximately 6-7% of patients remain severely symptomatic and require heart rate slowing agents. Other complaints such as decreased exercise capacity or effort dyspnea can occur in up to 14% of patients and they are usually attributed to faster than needed sinus rate at rest and during exercise.

Although in the vast majority of patients, the above mentioned symptoms are rather mild and do not decrease the patient's acceptance of CNA, in some may decrease the quality of life. Thus, a detailed assessment of the effects of CNA on exercise performance is clinically important. However, to date, no study addressed this issue.

There are several methods to assess exercise performance with cardiopulmonary exercise testing (CPET) being the most accurate and reference tool. It measures cardiorespiratory fitness and physiological responses to aerobic exercise in many conditions. CPET provides a comprehensive evaluation of the respiratory, circulatory, and metabolic responses to exercise that cannot be accurately measured by less precise methods such as standard exercise stress test. Therefore, we have chosen CPET to evaluate the effects of CNA on exercise performance in our patients.

Aim To assess one-year effects of CNA-induced total vagal denervation on cardiorespiratory fitness in patients undergoing CNA due to reflex asystolic syncope.

To compare cardiorespiratory fitness between subjects with reflex syncope and healthy volunteers.

Hypothesis. Cardioneuroablation significantly decreases cardiopulmonary fitness in patients with reflex asystolic syncope.

There are no differences between patients with syncope and healthy people in cardiorespiratory fitness at baseline whereas post-CNA results of CPET are significantly worse in syncope patients versus controls

Methods Patients. The study group will consist of consecutive patients undergoing CNA in our institution. Patients are referred for CNA if they have severe, recurrent symptoms due to reflex syncope with ECG documented asystole >3 seconds, especially if associated with injury, or recurrent presyncope with persistent reflex bradycardia. The patients have to have a history of ineffective prior non-pharmacological treatment and a positive baseline atropine test (sinus rate acceleration > 30% and no AV block following 2 mg of intravenous atropine). All patients gave informed written consent to undergo CNA and to participate in the study (Ethics Committee approval # 22/2024).

Control group. This group will consist of healthy volunteers without cardiovascular and other chronic disorders, age- and gender-matched with the CNA group. This group will not undergo CNA.

Cardioneuroablation. The procedure is performed under general anesthesia with muscle relaxation using a 3.5 mm irrigated tip catheter (Navistar ThermoCool SmartTouch) with contact force module and electroanatomical system Carto 3 (Biosense Webster, US). The ablation index is set at 500 except coronary sinus (CS) where the target value is 350. Intracardiac echocardiography (ICE) (Acuson SC2000, Siemens, Germany, AcuNav™ Ultrasound Catheter, Biosense Webster, US) is also used throughout the whole procedure and serves for guiding ablation, including identification of presumed GP areas. The extra cardiac vagal stimulation (ECVS) is performed using two diagnostic catheters positioned in the right and left jugular veins utilizing neurostimulator designed by Dr Pachon (Sao Paulo, Brazil) (pulse amplitude of 1 V/kg body weight up to 70 V, 50 ms width, 50 Hz frequency, delivered over 5 sec). Complete bilateral vagal denervation of both sinus and AV nodes (no sinus arrest, slowing of sinus rate no more than 10% compared with baseline and no AV block with PR interval no longer than at baseline), documented on ECVS, is the end-point of CNA.

Ablation is usually started in the left atrium (LA) at the anterior antrum of the right pulmonary vein where the superior paraseptal GP (SPSGP) is located, followed by ablation of the inferior paraseptal GP (IPSGP) at the floor of LA). Next, these GPs are ablated from the right atrium (RA). If the intraprocedural endpoints of CNA are not achieved by ablation of paraseptal GPs, additional applications in the LA at the sites of superior and postero-lateral LA GPs are performed, followed by applications in CS.

At the end of the procedure, atropine test is performed in order to assess the residual, if present, vagal nerve activity. The value of < 10% of increase in sinus rate following atropine injection (2 mg iv) will be taken as successful vagal denervation.

Cardiopulmonary exercise testing A symptom-limited cardiopulmonary exercise (CPET) will be performed twice, at baseline and after one year of follow-up, both in the syncope and control patients. Exercise tests will be performed on a treadmill with a cardio-pulmonary system Reynolds Medical. The same load protocol will be used twice for the same patient. All patients will be encouraged to exercise at maximal effort (≥8 points using the 10-point Borg scale). During the exercise test, the patient's clinical status will be monitored. The systolic and diastolic blood pressure will be recorded every 3 minutes of exercise. Heart rate, heart rate reserve (predicted and achieved), chronotropic index and percentage of maximum predicted heart rate at peak exercise will be calculated (3). The maximum predicted heart rate will be calculated as 220-age in years. The heart rate recovery in 1 minute will be assessed. A 12-lead electrocardiogram will be recorded. ECG and heart rate parameters: ischemia, arrhythmia, or conduction disturbances during exercise and recovery will be accessed according to the American Heart Association recommendations.

Ventilatory and gas exchange parameters will be assessed during the test. The peak oxygen uptake (VO2) will be averaged from the highest 30 s of exercise. Maximum predicted oxygen uptake will be calculated according to the Wasserman/Hansen equations. The anaerobic threshold will be calculated using a dual-method approach (V-slope and ventilatory equivalent methods). Other analyzed cardiopulmonary exercise testing parameters will include oxygen uptake to work rate increment ratio (∆O2/∆WR), ventilatory efficiency (VE/VCO2 slope), and breathing reserve at peak exercise, calculated as the percentage of maximum voluntary ventilation: [(maximum voluntary ventilation - minute ventilation at peak exercise) / maximum voluntary ventilation] × 100. All exercise tests will be supervised and analyzed according to current guidelines.

Quality of life. Quality of life will be measured using a dedicated questionnaire: The Impact of Syncope on Quality-of-Life Questionnaire University of Calgary. This questionnaire consists of 9 questions with 6 choices and 3 questions with 5 choices. The overall maximum score is 57. The higher the score the poorer the quality of life is.

Statistical analysis. The results are presented as mean±SD or numbers and percentages. Differences between variables are analysed using paired two-sided student t-test for normally distributed continuous variables or U Mann Whitney for not-normally distributed variables. The Chi square test (with Yates correction if appropriate) or exact Fisher test are used to compare qualitative parameters. A Pearson correlation coefficient is used to assess association between CPET values and QoL results. A p value < 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* severe, recurrent symptoms due to reflex syncope or recurrent presyncope due to slow heart rate
* ECG documented asystole >3 seconds
* ineffective prior non-pharmacological treatment
* positive baseline atropine test (sinus rate acceleration > 30% and no atrio-ventricular block following 2 mg of intravenous atropine)
* signed written informed consent

Exclusion Criteria:

* serious comorbidities precluding general anaesthesia and cardioneuroablation
* non-functional sinus arrest or atrio-ventricular block (negative atropine test)
* lack of consent to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
peak Vo2 | 12 months
  peak Vo2 = maximum amount of oxygen that body can absorb and use during exercise (ml/kg/min)

SECONDARY OUTCOMES:
chronotropic index | 12 months
  (peak heart rate-resting heart rate)/(220-age-resting heart rate) (%)
METs | 12 months
  metabolic equivalent of task (kcal/kg/min)
HR peak | 12 months
  maximal heart rate during exercise (beats/min)
HR reserve | 12 months
  heart rate reserve = the difference between peak heart rate during exercise and heart rate soon after stopping exercise.
exercise duration | 12 months
  duration of exercise in minutes and seconds
HR 1 minute after exercise | 12 months
  heart rate recorded one minute after completion exercise test (beats/min)

OTHER OUTCOMES:
Quality of Life | 12 months
  The Impact of Syncope on Quality-of-Life Questionnaire University of Calgary (points)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Piotrowski, PhD, Study Director — Department of Cardiology, Postgraduate Medical School, Grochowski Hospital
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
To share data on a reasonable request from other researchers in this filed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 24 months
Access Criteria: personal e-mail contact

REFERENCES:
- [Background] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Background] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276
- [Background] Piotrowski R, Baran J, Sikorska A, Krynski T, Kulakowski P. Cardioneuroablation for Reflex Syncope: Efficacy and Effects on Autonomic Cardiac Regulation-A Prospective Randomized Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):85-95. doi: 10.1016/j.jacep.2022.08.011. Epub 2022 Aug 28. PMID 36114133
- [Background] Kulakowski P, Baran J, Sikorska A, Krynski T, Niedzwiedz M, Soszynska M, Piotrowski R. Cardioneuroablation for reflex asystolic syncope: Mid-term safety, efficacy, and patient's acceptance. Heart Rhythm. 2024 Mar;21(3):282-291. doi: 10.1016/j.hrthm.2023.11.022. Epub 2023 Nov 29. PMID 38036236
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Rose MS, Koshman ML, Ritchie D, Sheldon R. The development and preliminary validation of a scale measuring the impact of syncope on quality of life. Europace. 2009 Oct;11(10):1369-74. doi: 10.1093/europace/eup106. PMID 19797151